CLINICAL TRIAL: NCT03082599
Title: Visual Outcomes of an Extended Depth of Focus (EDOF) Intraocular Lens (IOL)
Brief Title: Symfony Toric Intraocular Lens Visual Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other); Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 2016-002
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cataract Bilateral; Astigmatism Bilateral
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Emmetropia both eyes (OU) group (Active Comparator): Symfony Toric IOL target refraction both eyes emmetropia (±0.25D).
  Interventions: Device: Presbyopia and astigmatism correcting intraocular lens
- Nanovision group (Experimental): Symfony Toric IOL target refraction for the dominant eye will be plano (±0.25D) and for the non-dominant eye -0.50 ±0.16 D.
  Interventions: Device: Presbyopia and astigmatism correcting intraocular lens

INTERVENTIONS:
Device: Presbyopia and astigmatism correcting intraocular lens — The Symfony Toric IOL (ZXTx) is an extended depth of focus (EDOF) IOL design to improve the sharpness of vision at near, intermediate and far distances reducing the need of glasses after cataract surgery in patients with astigmatism.

SUMMARY:
In July 2016, the FDA approved an extended depth of focus (EDOF) IOL (Tecnis Symfony, Abbott Medical Optics) helping to improve the sharpness of vision at near, intermediate and far distances reducing the need of glasses after cataract surgery. It is available in both a non-toric version and a toric version for patients with astigmatism. The difference between this lens and the multifocal (MIOL) counterpart is that the EDOF, similarly to a monofocal IOL, has one focal point (elongated in the EDOF) while the multifocals have 2 focal points; therefore, having less of a halo and glare problem. Pivotal trial results where Symfony was compared to a monofocal IOL showed similar uncorrected distance visual acuity (UCDVA), better intermediate (77% vs. 34% 20/25 uncorrected intermediate visual acuity - UCIVA) and near vision (Symfony patients were able to read two additional, progressively smaller lines compared to the monofocal IOL).A One potential disadvantage of the EDOF IOL compared to a MIOL is the visual performance at near.B One option to deal with this potential shortcoming is to set the non-dominant eye for a small residual myopic error (-0.50 D)C what is referred to as nano-vision or mini mono-vision.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing bilateral cataract extraction with intraocular lens implantation.
2. Willing and able to provide written informed consent for participation in the study
3. Willing and able to comply with scheduled visits and other study procedures.
4. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6-15 days between surgeries.
5. Subjects who require an IOL power in the range of +5.0 D to +34.0 D only.
6. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Contact lens use during the active treatment portion of the trial.
5. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
6. Clinically significant corneal dystrophy
7. History of chronic intraocular inflammation.
8. History of retinal detachment.
9. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
10. Previous intraocular surgery.
11. Previous refractive surgery.
12. Previous keratoplasty
13. Severe dry eye
14. Pupil abnormalities
15. Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than yttrium aluminum garnet (YAG) capsulotomy, i.e. LASIK)
16. Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
17. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
18. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Study Chair — Carolina Eyecare Physicians, LLC
Locations (4):
- United States (4):
  - Associated Eye Care, Stillwater, Minnesota
  - Ophthalmic Consultants of Long Island, Garden City, New York
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Slade & Baker Vision Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 patients were enrolled and randomized; however, data from only 79 patients was analyzed due to major procedural issues at one site. One patient in the Emmetropia group missed the 3-month visit.
Period: Overall Study
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Started | 40 | 39
Completed | 39 | 39
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.1) | 69.0 (9.3) | 68.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 17 | 22 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 39 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 37 | 36 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance-corrected Near (40 cm) Visual Acuity.
Description: Visual acuity with correction (glasses) measured at 40 cm.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | 0.30 (0.14) | 0.26 (0.13)

2. Primary Outcome: Reduction of Manifest Cylinder (Diopters).
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | 1.15 (0.77) | 1.38 (0.80)

3. Secondary Outcome: Uncorrected Near (40 cm) Visual Acuity
Description: Visual acuity without correction (no glasses) measured at 40 cm.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | 0.25 (0.12) | 0.19 (0.12)

4. Secondary Outcome: Uncorrected Intermediate (66 cm) Visual Acuity
Description: Visual acuity without correction (no glasses) measured at 66 cm.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | 0.06 (0.10) | 0.04 (0.08)

5. Secondary Outcome: Uncorrected (4 m) Visual Acuity
Description: Visual acuity without correction (no glasses) measured at 4 m.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | -0.03 (0.08) | -0.02 (0.08)

6. Secondary Outcome: Modified Patient-Reported Visual Symptoms Questionnaire (PRVSQ)
Description: Percentage of patients who reported any visual symptoms such as halos, glare, starburst, light sensitivity when answering the self administered questionnaire.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
percentage of participants | 100 | 97.4

7. Secondary Outcome: Patient Reported Spectacle Independence Questionnaire
Description: Percentage of participants who reported wearing glasses none or a little of the time in the self administered questionnaire.
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
percentage of participants | 64.8 | 92.3

8. Other Pre Specified Outcome: Residual Mean Spherical Equivalent Refraction
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | -0.20 (0.22) | -0.33 (0.33)

9. Other Pre Specified Outcome: Residual Refractive Sphere
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | -0.30 (0.20) | -0.48 (0.37)

10. Other Pre Specified Outcome: Residual Refractive Cylinder
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
diopters | 0.20 (0.25) | 0.29 (0.27)

11. Other Pre Specified Outcome: Percentage of Eyes With Postoperative Manifest Refraction Spherical Equivalent (MRSE) Accuracy to Target ≤ 0.5D
Time Frame: 3 months
Population: One subject in the emmetropia group missed the Month 3 visit.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
Number analyzed (Participants) | 39 | 39
Number analyzed (Eyes) | 78 | 78
percentage of eyes | 100 | 88.4

ADVERSE EVENTS:
Time Frame: Average 3 months. Adverse events were collected from the moment patient enrolled in the study until exit.
Description: Only eye related events were collected.
Arm/Group | Emmetropia Both Eyes (OU) Group | Nanovision Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT03082599/Prot_SAP_000.pdf